CLINICAL TRIAL: NCT03308760
Title: Analytical and Functional Evaluation of Recovery Following Acute Rupture of the Achilles Tendon and Surgical Repair in Young Patients
Acronym: ACHILLE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GREMEAUX 2013
Record Dates: First submitted 2017-10-04; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Acute Unilateral Rupture of the Achilles Tendon
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Interview concerning the post-operative rehabilitation programme and a functional analysis using the American Orthopaedic Foot and Ankle Society questionnaire
Other: Static stabilometry — on a force plate, in a double- then single-foot stance, with the eyes open and then closed
Other: Isokinetic test — Isokinetic test of the flexors/extensors and invertors/evertors of the ankle

SUMMARY:
Acute rupture of the Achilles tendon is a very frequent sports injury. Surgical repair is the usual treatment in young subjects, and although the optimal technique is still a matter of debate, conventional surgery with a direct approach is still the reference technique in young sportsmen and women. Studies investigating the evolution of ankle muscle strength following surgery for a ruptured Achilles tendon are rare, even though it is a crucial criterion to determine the possibility of returning to the sport. This project thus proposes to study, in comparison with the healthy ankle:(1) the evolution of muscle strength in the flexors/extensors and invertors/evertors of the injured ankle, evaluated using an isokinetic dynamometer, and (2) the evolution of stabilometry parameters, at 6 months, then at 12 months, following surgery for acute unilateral rupture of the Achilles tendon, operated on using the conventional technique in young sportsmen and women and in comparison with the healthy side.

ELIGIBILITY:
Inclusion Criteria:

* persons informed about the research
* sportsmen and women (competition or leisure, practiced > 3h/week)
* Between 18 and 45 years old
* First episode of acute traumatic unilateral rupture of the Achilles tendon
* Open surgery in the Orthopaedic and Traumatology Department of Dijon University Hospital
* Identical post-operative immobilisation programme for 6 weeks
* Absence of major post-operative complications delaying the rehabilitation

Exclusion Criteria:

* persons without national health insurance cover
* concomitant joint disease that could be aggravated by the tests
* heart disease/contra-indication to effort required during the isokinetic test
* management other than open surgery (orthopaedic, functional, percutaneous surgery, …)
* Rupture of the contralateral tendon
* Contra-indication for the use of the Biodex S4 pro

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients followed at the Convalescence and Rehabilitation Unit of Dijon CHU
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 6 months
  measured on the healthy and injured side using an isokinetic dynamometer
Postural parameters measured using a stabilometry platform | 6 months
  measured using a stabilometry platform

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France